CLINICAL TRIAL: NCT03599947
Title: A Single-centre, Prospective Trial of the Detection of 5-hydroxymethylcytosine (5-hmC) in Plasma Cell-free DNA for Establishing a Model for the Early Diagnosis of Colorectal Cancer
Brief Title: A Model for the Early Diagnosis of Colorectal Cancer by the Detection of 5-hydroxymethylcytosine (5-hmC) in Plasma Cell-free DNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Prof., Fudan University
Other Study IDs: METHOD
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; early diagnosis; 5-hydroxymethylcytosine
MeSH Terms: conditions — Colorectal Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Peripheral venous blood

SUMMARY:
In this study, the investigators establish a model for the early diagnosis of colorectal cancer based on detection of 5-hydroxymethylcytosine (5-hmC) in training group and validate the effectiveness of the model using a validation group.

DETAILED DESCRIPTION:
Many kinds of cancers are associated with changes in epigenetics, including 5-methylcytosine (5-mC) and 5-hydroxymethylcytosine (5-hmC). This changes may help diagnose cancer. The new detection method for 5-hmC can meet the requirements of liquid biopsy.

The traditional diagnostic methods for colorectal cancer is colonoscopy and pathology which are inconvenient and unpleasant, and sometimes, it is difficult for the very patients to get tissues or get enough tissues. In addition, other screening methods for colorectal cancer,such as guaiac-based fecal occult blood testing and a blood test for methylated SEPT9 DNA, have the shortcomings of relatively low sensitivity and specificity. As a result, it is imperative to find a new detection method for early diagnosis of colorectal cancer with high the advantages of high sensitivity and specificity, minimally invasive and convenient.

The aim of this research study is to establish a model for the early diagnosis of colorectal cancer by the detection of 5-hmC in plasma cell-free DNA. Patients who are diagnosed with colorectal cancer by colonoscopy and pathology and not received any anti-tumor therapy (Arm A) will be eligible for inclusion as well as healthy individuals with normal colonoscopy (Arm B). Then, 5-hmC in plasma cell-free DNA will be detected and compared between the two arms of patients (training group) to establish a model to diagnosis other people (validation group) who may suffer from colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

Arm A

* Histologically proven colorectal adenocarcinoma
* No other malignancies in medical history except adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri
* Eastern cooperative oncology group score 0-2
* Informed consent

Arm B

* Healthy people with normal colonoscopy
* No other malignancies in medical history except adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri
* Eastern cooperative oncology group score 0-2
* Informed consent

Exclusion Criteria:

Arm A

* Patients received chemoradiotherapy or other anti-tumor therapy before being enrolled
* Patients and/or family members can not understand and accept this study
* Familial Adenomatosis Polyposis, Lynch Syndrome, acute inflammatory bowel disease
* Pregnancy or lactation
* Unsuitable to take part in the clinical trial judged by doctors

Arm B

* Pregnancy or lactation
* Unsuitable to take part in the clinical trial judged by doctors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with colorectal cancer or with normal colonoscopy.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2018-07-16 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the model in the diagnosis of colorectal cancer | 6-month
  Sensitivity and specificity of the model in the diagnosis of colorectal cancer in training group and validation group

CONTACTS AND LOCATIONS:
Locations (1):
- Wenju Chang, Shanghai, Shanghai Municipality, China